CLINICAL TRIAL: NCT06828666
Title: A Phase 1/2a, Multicenter, Randomized, Controlled, Single-Blind, Dose-Finding Study to Evaluate the Safety and Efficacy of Cryopreserved Devitalized Adipose Tissue Allograft (BRC-OA) for Pain Treatment in Subjects With Mild to Severe Osteoarthritis (OA) of the Knee
Brief Title: A Phase 1/2a to Evaluate the Safety and Efficacy of Adipose Tissue Allograft (BRC-OA) in Patients With Osteoarthritis of the Knee
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Britecyte (Network)
Collaborators: Amarex Clinical Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 241
Record Dates: First submitted 2025-02-05; First posted 2025-02-14 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-02

CONDITIONS: Osteoarthritis of Knee
Keywords: Pain Treatment in Osteoarthritis (OA) of the Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: The study will be conducted in two parts:
  * Part 1 (Safety Evaluation phase) - without control arm
  * Part 2 (Randomized Controlled phase) - with control arm
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part 1 - 2 mL of BRC-OA via intra-articular injection (Experimental)
  Interventions: Biological: Cryopreserved Devitalized Adipose Tissue Allograft
- Part 1 - 8 mL of BRC-OA via intra-articular injection (Experimental)
  Interventions: Biological: Cryopreserved Devitalized Adipose Tissue Allograft
- Part 2 - 2 mL of BRC-OA via intra-articular injection (Experimental)
  Interventions: Biological: Cryopreserved Devitalized Adipose Tissue Allograft
- Part 2 - 8 mL of BRC-OA via intra-articular injection (Experimental)
  Interventions: Biological: Cryopreserved Devitalized Adipose Tissue Allograft
- Part 2 - 2 mL of Normal Saline via intra-articular injection (Sham Comparator)
  Interventions: Other: Normal Saline (Placebo)

INTERVENTIONS:
Biological: Cryopreserved Devitalized Adipose Tissue Allograft — BRC-OA is a Cryopreserved Devitalized Adipose Tissue Allograft that has demonstrated anti-inflammatory and antioxidant properties of adipose tissue.
  Arms: Part 1 - 2 mL of BRC-OA via intra-articular injection; Part 1 - 8 mL of BRC-OA via intra-articular injection; Part 2 - 2 mL of BRC-OA via intra-articular injection; Part 2 - 8 mL of BRC-OA via intra-articular injection
Other: Normal Saline (Placebo) — 2 mL Normal Saline
  Arms: Part 2 - 2 mL of Normal Saline via intra-articular injection

SUMMARY:
The purpose of this study is to evaluate the safety profile of BRC-OA for pain treatment in patients with mild to severe OA of the knee, focusing particularly on two distinct doses. Alongside safety assessments, the study also aims to investigate the initial efficacy of BRC-OA in treating pain among these patients. The study product is a cryopreserved devitalized adipose tissue allograft (BRC-OA). BRC-OA is composed of a devitalized human adipose particulate that retains the inherent properties of adipose such as tissue architecture, extracellular matrix, and signaling molecules.

DETAILED DESCRIPTION:
The study will be conducted in two parts:

* Part 1 (Safety Evaluation phase) - without control arm
* Part 2 (Randomized Controlled phase) - with control arm

In Part 1, six subjects will be treated with a 7-day staggering interval between each subject's enrollment. The initial 3 subjects will receive a 2 mL dose of BRCOA, and if deemed safe and well-tolerated by the investigator, the next 3 subjects will receive an 8 mL dose, also following a 7-day staggering interval to assess safety and tolerability. Once both dose levels (2 mL and 8 mL) are confirmed to be safe and tolerable, the study will advance to Part 2. In Part 2, a total of 36 subjects (12 subjects per arm) will be randomized 1:1:1 to three parallel arms to be administered via intraarticular injection of 2 mL or 8 mL of BRC-OA, or 2 mL of normal saline (control).

ELIGIBILITY:
Inclusion Criteria:

1. Males or females 18-80 years of age, inclusive
2. Diagnosis of OA in one or both knees supported by documentation of clinical and radiographic findings(KL Grades 2-4) up to 6 months prior to screening:

   1. Diagnosis of degenerative or post-traumatic OA of the knee supported by documentation of clinical and radiographic findings up to 6 months prior to screening
   2. Degenerative meniscal tears allowed as long as there are no pending surgeries
   3. Flexion Contraction and Valgus/Varus deformity allowed if < 10 degrees
3. Subject must have tried for at least 3 months and failed on at least two of the following pharmacological standard of care therapies in the past 12 months:

   1. Acetaminophen
   2. NSAID (e.g., ibuprofen, naproxen)
   3. Opioid (e.g., tramadol)
   4. Topical NSAID (e.g., diclofenac gel)
   5. Intra-articular injections (e.g., corticosteroids, hyaluronic acid)
4. Subjects knee pain persists for at least 12 weeks prior to screening and does not improve with pain medications (e.g., NSAIDs, acetaminophen, tramadol, etc.) and/or other nonoperative treatment options
5. Index knee WOMAC pain subscale score of ≥ 40 on a normalized/standardized scale of 0 to 100 at screening visit Note: The index knee in subjects with bilateral OA of the knees is the one with worse pain with walking. Where both knees have equal pain with walking, then the knee on the subject's dominant side will be designated the index knee.

Exclusion Criteria:

1. BMI greater than 40 kg/m2
2. Previous IA injections (e.g., corticosteroid, hyaluronic acid (HA), platelet rich plasma (PRP), etc.) into the index knee within 3 months prior to screening
3. Prior Partial Joint Replacement (PJR) or Total Joint Replacement (TJR) of one or both knees
4. Knee surgery in the previous 6 months prior to enrollment and/or planned knee surgery during the study
5. Symptomatic OA of the hips, spine, or ankle that would interfere with the evaluation of the treated knee
6. Rapidly progressing osteoarthritis (RPOA)
7. Prior cartilage transplants in the index knee
8. Subjects who are actively treated with oral anticoagulants or heparin therapy (treatment such as low dose Aspirin and Plavix are allowed)
9. Current therapy with any immunosuppressive therapy, including corticosteroids (> 5mg/day of prednisone)
10. Any method of medical marijuana use containing THC or CBD, including smoke or vaporized spray inhalation, pills or liquids, edible foods, topical applications, etc.
11. Clinically significant intercurrent illness, medical condition, non-knee pain, or medical history that could jeopardize the patient safety, limit participation, or compromise interpretation of data derived from the patient; this includes neurological or mental illness, human immunodeficiency virus, fibromyalgia, complex regional pain syndrome, or any active infection - including hepatitis B or C
12. Active alcohol or substance use disorder, or any other reason that would make it unlikely for the patient to comply with study procedures
13. Females who are lactating or pregnant (positive pregnancy test for females of childbearing potential at screening Females of childbearing potential must be willing to use an acceptable method of contraception from screening up until 90 days after study drug injection administration Acceptable methods of contraception include abstinence, female subject/partner's use of hormonal contraceptive (oral, patch, injectable, depot, or vaginal) in conjunction with a barrier method (e.g., diaphragm, cervical cap, condom, spermicide, or sponge), or female subject/partner's use of an implantable device (implantable rod or intrauterine device)
14. Subject has known allergy to any components of BRC-OA
15. Subject has received an investigational product within 3 months before screening
16. Any medical condition, which in the opinion of the clinical investigator, would interfere with the treatment or outcome of the patient

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Outcome Measures | From Baseline to 6 months
  • Incidence and severity of local and systemic treatment-emergent adverse events (TEAEs) and SAEs
Primary Safety Outcome Measures | From Baseline to 6 months
  • Incidence of abnormal laboratory panel and vital signs (Baseline to 6 months)
Primary Efficacy Outcome Measure | From Baseline and 3 months
  • WOMAC VAS Pain Scale - WOMAC (Western Ontario and McMaster Universities Arthritis Index) pain subscale consists of 5 individual questions. The VAS score is determined by measuring in millimeters from the left-hand end of the line to the point that the patient marks (0-100 mm) for 5 questions [0 represents no knee pain, and 100 represents extreme knee pain]. The results for each question are summed to calculate the total WOMAC pain subscale score ranging from a total of 0 to 500. The total WOMAC pain subscale score will be normalized/standardized on a scale from 0 to 100. A negative number for the change from baseline indicates a reduction in pain.

SECONDARY OUTCOMES:
Secondary Efficacy Outcome Measures | Baseline to 6 months
  • WOMAC VAS Pain Scale - difference in change from Baseline and 1 week, 6 weeks, and 6 months
Secondary Efficacy Outcome Measures | Baseline to 6 months
  • WOMAC VAS Stiffness and Function Scales - difference in change from Baseline and 1 week, 6 weeks, 3 months, and 6 months
Secondary Efficacy Outcome Measures | Baseline to 6 months
  • WOMAC VAS Total Score - difference in change from Baseline and 1 week, 6 weeks, 3 months, and 6 months
Secondary Efficacy Outcome Measures | Baseline to 6 months
  • KOOS-12 Pain, Function, and Quality of Life Scales - difference in change from Baseline and 1 week, 6 weeks, 3 months, and 6 months
Secondary Efficacy Outcome Measures | Baseline to 6 months
  • KOOS-12 Summary Impact Score - difference in change from Baseline and 1 week, 6 weeks, 3 months, and 6 months
Secondary Efficacy Outcome Measures | Baseline and 3 months
  • SF-12 Questionnaire - difference in change from Baseline and 3 months
Secondary Efficacy Outcome Measures | Baseline to 6 months
  • Six-Minute Walk Test - difference in score from Baseline and 3 months and 6 months
Secondary Efficacy Outcome Measures | Baseline to 6 months
  • Rescue Treatments - percentage of subjects using rescue treatments from baseline to 1 week, 6 weeks, 3 months, and 6 months

OTHER OUTCOMES:
Additional Exploratory Outcome Measures | Baseline and 3 months
  • Inflammatory Biomarker Assessment (synovial fluid) - difference in change from Baseline and 3 months in inflammatory cytokine markers (e.g., IL-1, IL-6, TNF-α, etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Molly Saunders, Study Director — Sr. Director, Regenerative Medicine Programs
Locations (7):
- United States (7):
  - LifeBridge Health, Baltimore, Maryland
  - The Osteoporosis & Clinical Trials Center, Hagerstown, Maryland
  - MD Medical Research, Oxon Hill, Maryland
  - Elevate Clinical Research, Rockville, Maryland
  - Northwell Health, New York, New York
  - University Orthopedics Center, Altoona, Pennsylvania
  - University Orthopedics Center, State College, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided